CLINICAL TRIAL: NCT02558075
Title: Mood Lifters: A Self Help Program to Improve One's Psychological and Behavioral Well Being
Brief Title: Mood Lifters: A Self Help Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Patricia Deldin, Professor of Clinical Psychology, Associate Director of the University of Michigan Depression Center, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00097120
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Depression; Anxiety; Bipolar Disorder
MeSH Terms: conditions — Depression; Anxiety Disorders; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MoodLifters Program (Experimental): A program to provide evidence-based education and skills to reduce psychological distress and enrich people's lives.
  Interventions: Behavioral: MoodLifters Sessions

INTERVENTIONS:
Behavioral: MoodLifters Sessions — This program consists of 15 different sessions with a different topic for each session. These sessions will occur once a week for 15 weeks and will last approximately an hour each. These topics will be in one of five theoretically important areas: biological, cognitive, affective, behavioral and social. Each subsequent week will involve an in-depth exploration of each topic, including why it is important to mental well-being and practical ideas about how to implement positive changes into one's everyday life. Following the facilitator's brief presentation, group members will be invited to share their experiences, challenges, and provide peer support.

SUMMARY:
Large scale, effective, low-cost, and evidence-based programs that can nimbly translate new research discoveries into prevention and care for psychosocial based problems are urgently needed. This study hopes to provide support for Mood-Lifters, a template for a low-cost evidence based program, so that investigators may fill this gap and relieve suffering for millions of people who are not getting adequate mental health care. Mood-Lifters provides a low cost, research based program designed to enrich people's lives and reduce psychological distress. It is designed to provide useful support, coaching and information. It seeks to help people enhance pleasure, engagement and meaning in their lives while minimizing depression, fear, loneliness and other negative feelings via a proprietary peer based program that offers weekly meetings and other flexible support options. The goal of this pilot study is to test the efficacy of this program. This is not traditional therapy, rather an educational supportive program similar to WeightWatchers, but for mental health.

DETAILED DESCRIPTION:
Approximately half the population of the United States will meet criteria for a diagnosable mental illness over their lifetime. Many of these individuals will experience changes in productivity, family relationships and self-esteem. Some will engage in behaviors that endanger themselves or others. A small percentage of these people will receive treatment. This lack of treatment is partly due to stigma or lack of knowledge, but it is also due to lack of affordable or available services. Furthermore, even when people manage to receive care, it is often ineffective because it is not evidence-based.

This lack of prevention and treatment is costly. The economic burden of depression alone is second only to cardiovascular disease, and anxiety disorders cost the U.S. more than $42 billion per year. Moreover, it has been estimated that as many as 70% of primary care visits stem from psychosocial issues. This is problematic because primary care physicians often have neither the time nor expertise to provide adequate support for the wide range of psychosocial issues with which their patients are coping.

In short, a large scale, effective, low-cost, evidence-based program that can nimbly translate new research discoveries into prevention and care for psychosocial based problems is urgently needed. Mood Lifters intends to be the "Weight-watchers" of mental health and is a program designed to precisely fill these gaps and relieve these burdens for millions of people who are not getting adequate mental health care.

Weight watchers is a highly effective, evidence based, para-professionally delivered program that serves nearly 1.2 million customers a week. It serves a different population than a primary care physician or an obesity specialist. It is not bariatric surgery but rather supports the majority of people who need to lose weight. In comparison, Mood Lifters is not intensive psychiatric care. Rather, it serves an adjunctive service to primary care doctor's typical medical care (i.e., Medications) and utilizes a de-stigmatized service delivery model.

This study will pilot this innovative program. Researchers will test and refine the proof of concept in multiple community groups from Ann Arbor. Each group will consist of 8-12 participants who will be recruited from local communities via a variety of methods. Criteria for participation will be all adults who are not actively manic, suicidal or psychotic. These participants will not be able to participate and will be referred to mental health professionals.

This program consists of 15 different sessions with a different topic for each session. These sessions will occur once a week for 15 weeks and will last approximately an hour each. Prior to participation in the first session, participants will complete comprehensive baseline measures, including a comprehensive mood assessment and measures to assess their knowledge, attitudes, and behaviors relating to the topics to be covered. This will take approximately 2 hours. At each meeting, participants will complete a brief questionnaire on all the topics in order to track progress from week to week. Between weekly meetings, participants will practice and track their skill-building via a Daily & Weekly Points Checklist, which will include the topics discussed over the course of the program.

During the first group session, the group facilitator will provide an overview of the program, including the weekly topics. These topics will be in one of five theoretically important areas: biological, cognitive, affective, behavioral and social. Each subsequent week will involve an in-depth exploration of each topic, including why it is important to mental well-being and practical ideas about how to implement positive changes into one's everyday life. Following the facilitator's brief presentation, group members will be invited to share their experiences, challenges, and provide peer support.

At the conclusion of the program, each participant will again complete the comprehensive mood assessment as well as the same measures of knowledge, attitudes, and behaviors that were assessed at the beginning of the 15-week period. Additionally, participants will have the opportunity to complete these same measures at 1 month and 6 month post Mood Lifters program. A final analysis will then be conducted to assess the program's overall efficacy and its efficacy among the various populations described above. The results will be formally written up and reported, program modifications will be made, and further grant funding will be pursued.

ELIGIBILITY:
Exclusion Criteria:

* active suicidal thoughts or behavior
* active psychosis
* active mania.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction with Life Scale | 15 weeks post baseline assessment
  Change in overall satisfaction with life will be measured from baseline to 15 weeks.
Patient Health Questionnaire | 15 weeks post baseline assessment
  Change in depression symptomology will be measured from baseline to 15 weeks.
Generalized Anxiety Disorder scale | 15 weeks post baseline assessment
  Change in anxiety symptomology will be measured from baseline to 15 weeks.
Emotion visual analog scale | 15 weeks post baseline assessment
  change in emotion ratings (e.g. happy, sad, angry) will be measured on a visual analog scale ranging from not at all (happy, sad, angry) to extremely (happy, sad, angry).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gudzune KA, Bleich SN, Clark JM. Efficacy of Commercial Weight-Loss Programs. Ann Intern Med. 2015 Sep 1;163(5):399. doi: 10.7326/L15-5130-3. No abstract available. PMID 26322706
- [Background] Hattie JA, Sharpley CF, Rogers HJ. Comparative effectiveness of professional and paraprofessional helpers. Psychol Bull. 1984 May;95(3):534-41. No abstract available. PMID 6399757
- [Background] Patel V, Weiss HA, Chowdhary N, Naik S, Pednekar S, Chatterjee S, Bhat B, Araya R, King M, Simon G, Verdeli H, Kirkwood BR. Lay health worker led intervention for depressive and anxiety disorders in India: impact on clinical and disability outcomes over 12 months. Br J Psychiatry. 2011 Dec;199(6):459-66. doi: 10.1192/bjp.bp.111.092155. PMID 22130747